CLINICAL TRIAL: NCT07101393
Title: Determination of Postoperative Stroke Incidence in Patients With and Without the Use of Epiaortic Ultrasound in Coronary Artery Bypass Grafting Surgery
Brief Title: Postoperative Stroke and Epiaortic Ultrasound in CABG
Acronym: EAU and POCD
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ebubekir, PhD, Ataturk University
Other Study IDs: ES-01
Record Dates: First submitted 2025-07-13; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Delirium; Postoperative Stroke
Keywords: Epiaortic Ultrasound; Coronary Artery Bypass Grafting; Stroke; Postoperative Neurocognitive Impairment
MeSH Terms: conditions — Emergence Delirium; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EAU Use in CABG: This cohort includes patients who underwent isolated coronary artery bypass grafting (CABG) surgery between December 2023 and December 2024. The intervention group (EAU group) consisted of patients in whom epiaortic ultrasound (EAU) was used intraoperatively to assess atherosclerotic burden in the ascending and arch aorta. Findings from EAU guided intraoperative decision-making, including cannulation site and cross-clamp strategy. The control group comprised patients who underwent CABG without EAU. The primary outcomes evaluated were postoperative stroke incidence and neurocognitive impairment.
  Interventions: Procedure: Intraoperative Epiaortic Ultrasound (EAU)

INTERVENTIONS:
Procedure: Intraoperative Epiaortic Ultrasound (EAU) — Intraoperative epiaortic ultrasound (EAU) is a real-time imaging technique used during coronary artery bypass grafting (CABG) to evaluate the presence, location, and severity of atherosclerotic plaques in the ascending and arch aorta. In this study, EAU was performed after median sternotomy but prior to aortic manipulation, using a high-frequency linear transducer directly applied to the exposed aorta. Plaques were classified by thickness, and findings were used to guide surgical strategy, including modification of cannulation site, avoidance of cross-clamping, or alteration of grafting technique. This intervention differs from conventional CABG, in which such imaging is not routinely employed.
  Other Names: Epiaortic Scanning

SUMMARY:
This study aims to investigate the incidence of postoperative stroke and neurocognitive impairment in patients undergoing coronary artery bypass grafting (CABG), with or without the use of epi-aortic ultrasound (EAU). Atherosclerosis in the ascending aorta is a known risk factor for perioperative stroke and systemic embolization. The identification of atherosclerotic plaques before manipulation of the ascending aorta is important in minimizing embolic complications. Neurocognitive function will be assessed using the standardized Mini-Mental State Examination (SMMSE) before surgery and within 7 days postoperatively or at discharge. This prospective, observational, case-control study will evaluate the relationship between the presence of atherosclerotic plaques detected by EAU and neurocognitive and neurologic outcomes following CABG surgery.

DETAILED DESCRIPTION:
This is a prospective, observational case-control study designed to evaluate the association between the use of epi-aortic ultrasound (EAU) and the incidence of postoperative stroke and neurocognitive impairment following coronary artery bypass grafting (CABG) surgery. Patients undergoing elective CABG between December 2023 and December 2024 will be enrolled. Patients will be assigned to one of two groups based on the intraoperative use of EAU: the EAU group and the non-EAU group. EAU will be used to detect the presence, location, and characteristics of atherosclerotic plaques in the ascending aorta. Plaques will be categorized according to location and thickness (Stage 1-2: <3 mm, Stage 3-4-5: ≥3 mm). Neurocognitive function will be assessed preoperatively and postoperatively using the standardized Mini-Mental State Examination (SMMSE). Demographic variables and perioperative factors such as aortic cross-clamp time, cardiopulmonary bypass duration, and length of ICU stay will also be collected for analysis. The study aims to clarify the relationship between ascending aortic atherosclerosis detected by EAU and adverse neurological and cognitive outcomes, and to determine whether intraoperative EAU alters surgical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for isolated, elective coronary artery bypass grafting (CABG)
* Age 18 years or older

Exclusion Criteria:

* Illiteracy (inability to read or write)
* Visual and/or hearing impairment
* Non-citizens/foreign nationals
* Refusal to participate in the study
* Presence of neuropsychiatric disorders that may affect postoperative cognitive evaluation (e.g., psychosis, dementia, mental retardation)
* History of cerebrovascular accident (CVA/stroke)
* Preoperative rhythm disturbances associated with stroke risk (e.g., atrial fibrillation, atrial flutter)
* Presence of intracardiac thrombus (ventricular or atrial) on preoperative echocardiography
* Patients undergoing concomitant cardiac procedures (e.g., valve or aortic surgery)
* Emergency CABG surgery
* Recent myocardial infarction
* Use of intra-aortic balloon pump (IABP)
* Redo CABG surgery
* Significant carotid stenosis or plaque detected on preoperative carotid Doppler ultrasonography
* Chronic renal failure and/or liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged ≥18 years) who underwent isolated, elective coronary artery bypass grafting (CABG) surgery at a single cardiovascular surgery center between December 2023 and December 2024. All participants were evaluated preoperatively for eligibility based on cognitive and clinical criteria. Patients were assigned to either the intervention group (with intraoperative epiaortic ultrasound use) or the control group (without EAU use). Individuals with neuropsychiatric disorders, prior stroke, rhythm disturbances, or other major comorbidities were excluded to ensure reliable neurocognitive assessment.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Stroke | Within 10 days postoperatively
  Occurrence of new-onset ischemic stroke confirmed by clinical neurological evaluation and neuroimaging (CT or MRI) within 10 days following coronary artery bypass grafting (CABG) surgery.

SECONDARY OUTCOMES:
Postoperative Neurocognitive Impairment (PNCI) | Up to 7 days postoperatively or at hospital discharge
  Neurocognitive status was assessed using the Standardized Mini-Mental State Examination (SMMSE), which ranges from 0 to 30, with higher scores indicating better cognitive function. A score of <20 was defined as clinically significant neurocognitive impairment. Evaluations were performed preoperatively and repeated at discharge or within 7 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: ebubekir sonmez, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made publicly available due to institutional policies and the potential for overlapping use of the same dataset by other researchers within the institution. However, data may be shared upon reasonable request, provided that appropriate ethical approvals and data-sharing agreements are in place

REFERENCES:
- [Result] Shapeton AD, Leissner KB, Zorca SM, Amirfarzan H, Stock EM, Biswas K, Haime M, Srinivasa V, Quin JA, Zenati MA. Epiaortic Ultrasound for Assessment of Intraluminal Atheroma; Insights from the REGROUP Trial. J Cardiothorac Vasc Anesth. 2020 Mar;34(3):726-732. doi: 10.1053/j.jvca.2019.10.053. Epub 2019 Nov 9. PMID 31787434

DOCUMENTS (1):
  • Informed Consent Form (2025-07-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT07101393/ICF_000.pdf